CLINICAL TRIAL: NCT02316912
Title: Double Blind Randomised Placebo Controlled Evaluation of Single and Multiple Oral Doses of ATX2417 in Man and Effect of Food
Brief Title: First in Man Evaluation of Single and Multiple Doses of Oral ATX2417
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atopix Therapeutics, Ltd. (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: ATX2417/001/14
Record Dates: First submitted 2014-12-02; First posted 2014-12-15 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Allergy
Keywords: allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (18):
- Single dose level 1 active (Active Comparator): Six subjects ATX2417 I mg tablet once.
  Interventions: Drug: ATX2417
- Single dose level 2 active (Active Comparator): Six subjects ATX2417 2x1 mg tablet once.
  Interventions: Drug: ATX2417
- Single dose level 3 active (Active Comparator): Six subjects ATX2417 5 mg tablet once.
  Interventions: Drug: ATX2417
- Single dose level 4 active (Active Comparator): Six subjects ATX2417 4x5 mg tablets once.
  Interventions: Drug: ATX2417
- Single dose level 5 active (Active Comparator): Six subjects ATX2417 to be determined.
  Interventions: Drug: ATX2417
- Multiple dose level 1 active (Active Comparator): Six subjects ATX2417 dose to be determined once daily for 8 days.
  Interventions: Drug: ATX2417
- Multiple dose level 2 active (Active Comparator): Six subjects ATX2417 dose to be determined once daily for 8 days.
  Interventions: Drug: ATX2417
- Single dose level 1 placebo (Placebo Comparator): Two subjects one placebo tablet once.
  Interventions: Drug: Placebo
- Single dose level 2 placebo (Placebo Comparator): Two subjects one placebo tablet x2 once.
  Interventions: Drug: Placebo
- Single dose level 3 placebo (Placebo Comparator): Two subjects one placebo tablet once.
  Interventions: Drug: Placebo
- Single dose level 4 placebo (Placebo Comparator): Two subjects two placebo tablets once.
  Interventions: Drug: Placebo
- Single dose level 5 placebo (Placebo Comparator): Two subjects four placebo tablets once.
  Interventions: Drug: Placebo
- Multiple dose level 1 placebo (Placebo Comparator): Two subjects matching placebo(s) once daily for 8 days
  Interventions: Drug: Placebo
- Multiple dose level 2 placebo (Placebo Comparator): Two subjects matching placebo(s) once daily for 8 days.
  Interventions: Drug: Placebo
- Single dose level 6 active (Active Comparator): Six subjects ATX2417 to be determined.
  Interventions: Drug: ATX2417
- Single dose level 7 active (Active Comparator): Six subjects ATX2417 to be determined.
  Interventions: Drug: ATX2417
- Single dose level 6 placebo (Placebo Comparator): Six subjects placeboto be determined.
  Interventions: Drug: Placebo
- Single dose level 7 placebo (Placebo Comparator): Six subjects placebo to be determined.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ATX2417 — Randomised double blind parallel group ascending dose assessment
  Arms: Multiple dose level 1 active; Multiple dose level 2 active; Single dose level 1 active; Single dose level 2 active; Single dose level 3 active; Single dose level 4 active; Single dose level 5 active; Single dose level 6 active; Single dose level 7 active
Drug: Placebo — Randomised double blind parallel group ascending dose assessment
  Arms: Multiple dose level 1 placebo; Multiple dose level 2 placebo; Single dose level 1 placebo; Single dose level 2 placebo; Single dose level 3 placebo; Single dose level 4 placebo; Single dose level 5 placebo; Single dose level 6 placebo; Single dose level 7 placebo

SUMMARY:
First in man evaluation of single and multiple doses of compound ATX2417 in healthy male volunteers. A double blind placebo controlled parallel group ascending dose design; up to five dose levels for the single dose and up to two dose levels for the multiple dose (8 days of dosing). Subjects will be screened to assure normal health prior to inclusion in the trial and will be monitored for safety (adverse events, vital signs, ECGs, safety labs) and pharmacokinetic profile. A fasted/fed comparison will also be included in the single ascending dose part of the trial.

DETAILED DESCRIPTION:
The study consists of two parts, A (single ascending dose including fasted/fed comparison) and B (multiple ascending dose). Part B will be conducted after a thorough review by the Sponsor and the Principal Investigator of the data arising from part A.

Part A This will be a randomised, double blind, placebo controlled, parallel group titration of up to seven single dose levels of ATX2417. In each cohort, six subjects will receive active compound and two will receive placebo in a randomised fashion. At each dose level, 2 subjects (1 subject will receive ATX2417 and 1 subject will receive placebo) will be dosed on Day 1 and the remaining 6 subjects will be dosed at least 24 hours later. Safety and pharmacokinetic observations will be made. There will be a minimum of two weeks between the first dosing day at each dose level. Safety and ATX2417 pharmacokinetic data will be reviewed prior to each dose escalation and, based on pharmacokinetic data, it is also possible to decrease the dose if the pharmacokinetic profile so indicates. This part will also include an assessment of the effect of a high fat breakfast on the absorption and pharmacokinetic profile of ATX 2417, performed at a dose predicted to be associated with therapeutic plasma concentrations.

Part B Following completion of Part A, and selection of appropriate dose levels, Part B will be performed. This will be a randomised, double blind, placebo controlled, parallel group study of up to two dose levels of ATX2417 given once daily for eight days. In each cohort, six subjects will receive active compound and two will receive placebo in a randomised fashion. Safety and pharmacokinetic observations will be made.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects, any racial group
2. Able to comply with the protocol
3. Subjects with a Body Mass Index (BMI) of 21-28 (BMI = Body weight (kg) / (Height (m)2)

Exclusion Criteria:

1. A history of gastrointestinal disorder likely to influence drug absorption
2. Receipt of any medication including over the counter preparations and vitamins within 14 days of the first dose of study drug with the exception of paracetamol up to a maximum of 2 g daily
3. Evidence of clinically significant renal, hepatic, cardiovascular or metabolic dysfunction
4. A history of drug or alcohol abuse
5. Inability to communicate well with the investigator (i.e., language problem, poor mental development or impaired cerebral function)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2015-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events as a measure of safety and tolerability | 120 hours after dosing
  Number of subjects with adverse events

SECONDARY OUTCOMES:
AUC0-t | 120 hours after single dose
  Area under concentration time curve at 120 hours
AUC0-t | 120 hours after eighth dose
  Area under concentration time curve at 120 hours

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Abou Farha, MD, Principal Investigator — Simbec Research
Locations (1):
- Simbec Research, Merthyr Tydfil, Glamorgan, United Kingdom